CLINICAL TRIAL: NCT02901392
Title: Fundación Instituto Valenciano de Oncología Prospective Registry for Patients Undergoing Male Sling or Artificial Urinary Sphincter After Prostatectomy or Radiation Therapy for Prostate Cancer.
Brief Title: Fundación IVO Registry for Patients Undergoing Sling or Artificial Urinary Sphincter After Prostate Cancer Treatment
Status: Recruiting | Type: Observational
Sponsor: Fundación Instituto Valenciano de Oncología (Other)
Responsible Party: Sponsor
Other Study IDs: Oncodinamia01
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2018-08-02 (Actual); Status verified 2018-07

CONDITIONS: Urinary Incontinence, Stress
Keywords: Male Urethral Slings; Artificial Urinary Sphincter; Prostatectomy; Radiotherapy
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 15 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Artificial urinary sphincter AMS-800®: Male patients with stress urinary incontinence after prostatectomy or radiotherapy treated with AMS-800®
  Interventions: Procedure: AMS-800
- AdVance/AdvanceXP®: Male patients with stress urinary incontinence after prostatectomy or radiotherapy treated with AdVance/AdvanceXP®
  Interventions: Procedure: ADVANCE/ADVANCEXP
- VIRTUE®: Male patients with stress urinary incontinence after prostatectomy or radiotherapy treated with VIRTUE®
  Interventions: Procedure: VIRTUE
- INVANCE®: Male patients with stress urinary incontinence after prostatectomy or radiotherapy treated with INVANCE®
  Interventions: Procedure: INVANCE

INTERVENTIONS:
Procedure: AMS-800 — Artificial urianry sphincter
  Groups: Artificial urinary sphincter AMS-800®
Procedure: ADVANCE/ADVANCEXP — Male sling
  Groups: AdVance/AdvanceXP®
Procedure: VIRTUE — Male sling
  Groups: VIRTUE®
Procedure: INVANCE — Male sling
  Groups: INVANCE®

SUMMARY:
Stress urinary incontinence is a significant potential source of morbidity after radical prostatectomy or radiation therapy for prostate cancer. At present, artificial urinary sphincter remains the preferred therapeutic option. However, this technique is not free from complications. In an attempt to avoid such complications, male sling has been suggested for use in patients with mild degrees of stress incontinence.

DETAILED DESCRIPTION:
This is a prospective collection of pre-defined parameters on the treatment of male stress urinary incontinence by male sling or artificial urinary sphincter.

This registry includes:

1. Pre-operative urodynamic assessment, cystoscopy and other preoperative clinical parameters (i.e. age, body mass index, bladder neck contracture treated, urgency, 24h-PW, cystometry and pressure/flow, repositioning test)
2. Description of surgical technique
3. Continence is evaluated 3 months after surgery, avoiding the potential confounding impact of the initial tissue edema (Cure was defined as no pad use, and all other cases were defined as failures)
4. Evaluation of long term functional outcome (efficacy, late complications and the loss of continence)

Surgery is performed with:

Device: Virtue® Device: Advance® and AdvanceXP® Device: Artificial urinary sphincter AMS-800® Device: Invance® Male Incontinence Sling

A prospective functional follow-up, with 24h-Pad Weight test and ICIQ-UI SF, is carried out 3-monthly for the first year and 6-monthly thereafter, parallel to the oncological follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. The subject has agreed to be treated with the male Incontinence surgery devices
2. The subject is willing and able to give valid informed consent.
3. The subject is > 18 years of age.
4. The subject has confirmed stress urinary incontinence for at least 12 months after prostatectomy or radiotherapy.
5. It has been confirmed the stress urinary incontinence with 24-Hour Pad Weight test
6. Pre-operative urodynamic assessment and flexible cystoscopy were performed in all cases
7. The subject is willing and able to return for follow-up evaluations and questionnaire completion according to the study protocol.
8. There are no surgical contraindications.

Exclusion Criteria:

1. The subject has an active urinary tract infection or active skin infection in region of surgery
2. The subject has serious bleeding disorders
3. The subject has unstable bladder neck stricture disease
4. The subject has Neurogenic bladder condition that is not treatable or controllable by pharmacological or alternative methods.
5. The subject has Detrusor-external sphincter dyssynergia.
6. The subject is unable or unwilling to sign the informed consent form (ICF)and/or comply with all follow-up requirements according to the study protocol
7. The subject is likely to undergo radiation therapy within the next 6 months
8. The subject has a history of connective tissue or autoimmune conditions.
9. The subject has a compromised immune system.
10. The subject has renal insufficiency, and upper and/or lower urinary tract relative obstruction.
11. The subject's reading level is judged inadequate for reading and understanding the quality of life questionnaires and other study materials

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stress urianry incontinence undergoing male sling or artificial urinary sphincter after prostatectomy or radiation therapy for prostate cancer
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2004-04; Primary Completion 2019-04 (Estimated); Study Completion 2031-04 (Estimated)

PRIMARY OUTCOMES:
Success rate | 3 months
  Cure is defined as no pad use

SECONDARY OUTCOMES:
Continence improvement | 15 years
  Assessed by means of the 24-Hour Pad Weight test
Lower tract urinary symptoms modification after male surgery incontinence | 15 years
  Assessed with IPSS questionaires
Quality of Life in patients with male surgery incontinence | 15 years
  Assessed with "International Consultation on Incontinence Questionnaire -- Short Form (ICIQ-SF)" questionaires

CONTACTS AND LOCATIONS:
Overall Officials: Argimiro Collado, MD,PhD, Principal Investigator — Fundación IVO
Locations (1):
- Argimiro Collado, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Collado A, Gomez-Ferrer A, Rubio-Briones J, Bonillo MA, Iborra I, Solsona E. [Which patients with stress urinary incontinence after radical prostatectomy benefit from the indication of an Invance?]. Arch Esp Urol. 2009 Dec;62(10):851-9. doi: 10.4321/s0004-06142009001000010. Spanish. PMID 20065535
- [Result] Collado Serra A, Resel Folkersma L, Dominguez-Escrig JL, Gomez-Ferrer A, Rubio-Briones J, Solsona Narbon E. AdVance/AdVance XP transobturator male slings: preoperative degree of incontinence as predictor of surgical outcome. Urology. 2013 May;81(5):1034-9. doi: 10.1016/j.urology.2013.01.007. Epub 2013 Mar 7. PMID 23465151
- [Result] Collado Serra A, Dominguez-Escrig J, Gomez-Ferrer A, Batista Miranda E, Rubio-Briones J, Solsona Narbon E. Prospective follow-up study of artificial urinary sphincter placement preserving the bulbospongiosus muscle. Neurourol Urodyn. 2017 Jun;36(5):1387-1394. doi: 10.1002/nau.23119. Epub 2016 Sep 21. PMID 27654121
- [Result] Collado A, Dominguez-Escrig J, Ortiz Rodriguez IM, Ramirez-Backhaus M, Rodriguez Torreblanca C, Rubio-Briones J. Functional follow-up after Advance(R) and Advance XP(R) male sling surgery: assessment of predictive factors. World J Urol. 2019 Jan;37(1):195-200. doi: 10.1007/s00345-018-2357-9. Epub 2018 Jun 8. PMID 29948042